CLINICAL TRIAL: NCT04321083
Title: Measurement of Cerebral rSO2 Levels During Sleep in Children With Suspected Obstructive Sleep Apnea
Acronym: O2SLEEP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC18AD078918CTIL
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea; Pediatric Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: INVOS Medtronic device will be applied simultaneously with sleep lab monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes

ARMS (1):
- O2 brain (central) measurement (Experimental): INVOS will be applied simultaneously for monitoring along with the regular polysomnography (sleep lab) workup
  Interventions: Diagnostic Test: INVOS

INTERVENTIONS:
Diagnostic Test: INVOS — INVOS monitoring brain o2 saturation

SUMMARY:
The gold standard of obstructive sleep apnea (OSA) is (PSG)POLYSOMNOGRAPHY. During the examination, the patient is monitored by saturation, EEG and other measurements.

Near infrared spectroscopy is an uprising technology allowing non invasive measurement of the frontal lobe oxygenation. It is painless and does not have side effects. We believe that brain saturation will be more accurate then peripheral pulse oximeter and will be better correlated with the clinical presentation of OSA.

DETAILED DESCRIPTION:
a prospective cohort study study group - pediatric population referred to PSG in Dana Duek Hospital. After informed consent received from the parents, the parents will fulfill "Connors" (age 6 +) & "Brief" (age 4-6) questionnaires.

During the PSG, the brain saturation will be monitored by INVOS(TM) Medtronic device. They will be monitored & synchronized with the peripheral saturation documented performed as part of the PSG examination.

The brain saturation & peripheral saturation levels will be compared and both will be correlated to the questionnaires & AHI.

ELIGIBILITY:
Inclusion Criteria:

* 4-16 y/o pediatric population referred for PSG in Dana Hospital

Exclusion Criteria:

* down synd.
* craniofacial malformation
* PPD

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation between brain o2 levels to peripheral measurements | procedure (during the examination PGS)
  correlation between brain o2 levels to peripheral measurements

CONTACTS AND LOCATIONS:
Overall Officials: Ari Derowe, prof, Principal Investigator — Dana Duek pediatric hospital, TASMC, TA, ISRAEL
Locations (1):
- Dana Duek pediatric hospital TASMC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No